CLINICAL TRIAL: NCT04031989
Title: Phase Signal Acquisition System (PSAQ): Repository of Phase Signals for Pulmonary Hypertension Algorithm Development
Brief Title: Repository of Phase Signals for Pulmonary Hypertension Algorithm Development
Acronym: IDENTIFY - PH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Analytics For Life (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHDEV-CIP-001
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Right Heart Failure; Cardiac Disease
Keywords: Pulmonary Hypertension; Right Heart Cath
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Heart Diseases; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Repository study designed to collect signals using the CorVista Capture in subjects scheduled for Right Heart Catheterization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Enrolled Subjects (PSR) (Other): Patients who meet the study's entrance criteria and provide written informed consent, will undergo signal acquisition prior to their scheduled right heart catheterization (RHC) on the day of the procedure.
  Interventions: Device: CorVista Capture

INTERVENTIONS:
Device: CorVista Capture — The CorVista System is a medical device system that is being developed to collect phase signals from patients to support the development and testing of machine learned algorithms developed by CorVista Health. Data collected with the CorVista System during this study will not be used to guide treatment.

SUMMARY:
This study is designed as a repository study to collect resting cardiac phase signals and subject meta data from eligible subjects using the Phase Signal Recorder (PSR) prior to Right Heart Cath (RHC). The repository data will be used for the purposes of research, development, optimization and testing of machine-learning algorithms developed by CorVista Health (formerly Analytics 4 Life).

DETAILED DESCRIPTION:
Male and Female subjects will be uniquely and consecutively enrolled into one group to support populating a repository of phase signals. Resting phase signals will be collected in all patients who meet inclusion/exclusion criteria and have signed an informed consent form. This study consists of a screening visit, resting phase signal collection (study procedure), and right heart catheterization. In this study, resting phase signals will be acquired in subjects prior to Right Heart Catheterization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old;
2. Scheduled to undergo right heart catheterization;
3. Ability to understand the requirements of the study and to provide written informed consent.
4. Normal Sinus Rhythm (SSR) at time of phase signal collection.

Exclusion Criteria:

1. Prior heart valve replacement
2. Prior lung or heart transplant
3. Infiltrative myocardial disease (amyloid, sarcoid, right ventricular dysplasia);
4. Presence of cardiac implantable electronic device (CIED), including implantable cardioverter defibrillator (ICD), pacemaker (PM), implantable loop recorders and other monitors;
5. Implantable Neuro-stimulators;
6. Congenital Heart Disease;
7. Pregnant or breast feeding;
8. Currently taking any Type IA, IC or III antiarrhythmics;
9. Any history of amiodarone use;
10. Clinically significant chest deformity (e.g., pectus excavatum or pectus carinatum);
11. Breast implants;
12. Neuromuscular Disease if the condition results in tremor or muscle fasciculations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Phase Signal Recorder Procedure | 7 day
  Resting phase signals will be collected from eligible subjects prior to Right Heart Catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Horace R Gillins, BS CCRP, Study Director — CorVista Health; William E Sanders, Jr, MD JD LLM MBA FHRS, Study Director — CorVista Health
Locations (17):
- United States (17):
  - UC-MHS (UCHealth Memorial), Colorado Springs, Colorado
  - University of Colorado-MHS (UCHealth Memorial), Colorado Springs, Colorado
  - WellStar Research Institute, Marietta, Georgia
  - Loyola University Chicago, Maywood, Illinois
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Bryan Heart, Lincoln, Nebraska
  - The Rochester General Hospital, Rochester, New York
  - Duke University, Durham, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Allegheny Health Network Research Institute, Natrona Heights, Pennsylvania
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Lexington Cardiology / Lexington Medical Heart and Vascular Center, Lexington, South Carolina
  - Austin Heart, Austin, Texas
  - Sentara Hospitals and Sentara Medical Group, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No